CLINICAL TRIAL: NCT04870632
Title: Six Weeks Tele-based Resistance Exercise Improves the Respiratory Muscle Strength and Biceps Strength Among Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Tele-based Resisted Exercise for COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Ching-Hsia Hung, Professor, National Cheng-Kung University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-108-038-2
Record Dates: First submitted 2021-04-14; First posted 2021-05-03 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: COPD; Pulmonary Rehabilitation; Telerehabilitation; Cardiopulmonary Exercise Test; Compliance, Patient
Keywords: COPD; Pulmonary Rehabilitation; Telerehabilitation; Video-based telerehabilitation; Youtube; LINE; Booklet-based telerehabilitation; Cardiopulmonary exercise test; Interval strengthening exercises; Cellphone
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Compliance | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Sham Comparator): Patients in control group received the education booklet with words and pictures.
  Interventions: Other: Education
- Video group (Experimental): Patients in intervention group watched YOUTUBE videos to rehab and recorded the intensity after the exercise by RPE scores. During the intervention, a physical therapist would have weekly telephone calls or LINE calls for 6 times to monitor and modify the intensity of exercise.
  Interventions: Other: Video-based pulmonary rehabilitation
- Booklet group (Experimental): Patients in intervention group read education booklet with words and pictures to rehab and recorded the intensity after the exercise by RPE scores. During the intervention, a physical therapist would have weekly telephone calls or LINE calls for 6 times to monitor and modify the intensity of exercise.
  Interventions: Other: Booklet-based pulmonary rehabilitation

INTERVENTIONS:
Other: Education — COPD patients conduct pulmonary rehabilitation for 6 weeks by read an education booklet with words and pictures which is made by the physiotherapist.
  Arms: Control group
Other: Video-based pulmonary rehabilitation — COPD patients conduct pulmonary rehabilitation for 6 weeks by watching Youtube videos which were made by the physiotherapist.The patients are monitored by the physiotherapist by weekly phone call and asked to record RPE scores at the RPE form.
  Arms: Video group
Other: Booklet-based pulmonary rehabilitation — COPD patients conduct pulmonary rehabilitation for 6 weeks by read an education booklet with words and pictures which is made by the physiotherapist.The patients are monitored by the physiotherapist by weekly phone call and asked to record RPE scores at the RPE form.
  Arms: Booklet group

SUMMARY:
The present study aims to investigate the effect of six weeks tele-based resisted exercises on cardiopulmonary function, quality of life, muscle strength and functioanl performance among patients with chronic obstructive pulmonary disease. In addition, the effect of different forms of exercise instruction (i.e., booklet and video) was also investigated.

DETAILED DESCRIPTION:
Background and Purpose: Chronic obstructive pulmonary disease (COPD) is the 3rd global cause of deaths. Pulmonary rehabilitation (PR) is the standard treatment for this disease. However, the dropout rate remains high (33-50%) because of traffic issues and patients' low mobility. Therefore, telerehabilitation seems to be a better way to deliver PR. Using videos to deliver PR is not only easy to manipulate on the cellphone or ipad, but also improve patients' attention and compliance. Thus, the aim of this study is to assess whether tailor-made PR video rehabilitation program improves patients' quality of life (QoL), muscle strengths, cardiopulmonary functions, and compliance.

Methods: This is a quasi-experimental study. Participants were medically stable COPD patients and able to use LINE and YOUTUBE in cellphone. They voluntarily choose to participate in control group, booklet group or video groups to conduct 6-week tele-based resisted exercise program. Patients in control group received conventional intervention and exercise instruction booklet. Participants in booklet and video groups additionally received a COPD exercise package with 2 elastic bands in different weight (4 ponds and 8 ponds). Participants in booklet group received the exercise instructed in education booklet with words and pictures. Patients in video group received exercise instructed using YouTube videos. Both participants in booklet and video groups were asked to record their rating of perceived exertion (RPE) scores. A physical therapist would weekly contact them to monitor and modify the exercise intensity using their RPE scores. The videos included 5-minute breathing reeducation, 20-minute interval strengthening exercise and 5-minute education animation. All patients were assessed the performance of spirometry, cardiopulmonary exercise test (CPET), questionnaires about symptoms, QoL, muscle strengths and distances of 6-minute walk test (6MWT) before intervention, after intervention and after 6-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Be medically stable
* Ability to use a smartphone and applications (LINE and Youtube)
* Access to the internet
* Have visual and auditory impairments corrected with assistive devices

Exclusion Criteria:

* Other respiratory disease as main complaint other than COPD
* Exacerbations within 4 weeks
* Had enrolled PR programs within the last 6 months
* Unable to follow verbal instructions, suffer from cognitive impairment, or have language difficulties
* Unstable medical conditions
* Any comorbidities which precluded exercise training

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Time point difference of AT from 1st week to 6th week | From 1st week to 6th week
  Use cardiopulmonary exercise test (CPET) to get the change of time point difference of AT from 1st week(intervention starts) to 6th week(intervention ends)
Time point difference of AT from 1st week to 12th week | From 1st week to 12th week
  Use cardiopulmonary exercise test (CPET) to get the change of time point difference of AT from 1st week(intervention starts) to 12th week(follow up ends)
Time point difference of AT from 6th week to 12th week | From 6th week to 12th week
  Use cardiopulmonary exercise test (CPET) to get the change of time point of AT from 6th week(intervention ends) to 12th week(follow up ends)
Change of maximal exercise work from 1st week to 6th week | From 1st week to 6th week
  Use cardiopulmonary exercise test (CPET) to get the change of values of the pateint's total work (watt) from 1st week(intervention starts) to 6th week(intervention ends)
Change of maximal exercise work from 1st week to 12th week | From 1st week to 12th week
  Use cardiopulmonary exercise test (CPET) to get the change of values of the pateint's total work (watt) from 1st week(intervention starts) to to 12th week(follow up ends)
Change of maximal exercise work from 6th week to 12th week | From 6th week to 12th week
  Use cardiopulmonary exercise test (CPET) to get the change of values of the pateint's total work (watt) from 6th week(intervention ends) to 12th week(follow up ends)
Change of VO2max from 1st week to 6th week | From 1st week to 6th week
  Use cardiopulmonary exercise test (CPET) to get the change of values of VO2max (mL/min/kg) from 1st week(intervention starts) to 6th week(intervention ends)
Change of VO2max from 1st week to 12th week | From 1st week to 12th week
  Use cardiopulmonary exercise test (CPET) to get the change of values of VO2max (mL/min/kg) from 1st week(intervention starts) to 12th week(follow up ends)
Change of VO2max from 6th week to 12th week | From 6th week to 12th week
  Use cardiopulmonary exercise test (CPET) to get the change of values of VO2max (mL/min/kg) from 6th week(intervention ends) to 12th week(follow up ends)
Change of VE/VCO2 from 1st week to 6th week | From 1st week to 6th week
  Use cardiopulmonary exercise test (CPET) to get the change of values of VE/VCO2 from 1st week(intervention starts) to 6th week(intervention ends)
Change of VE/VCO2 from 1st week to 12th week | From 1st week to 12th week
  Use cardiopulmonary exercise test (CPET) to get the change of values of VE/VCO2 from 1st week(intervention starts) to 12th week(follow up ends)
Change of VE/VCO2 from 6th week to 12th week | From 6th week to 12th week
  Use cardiopulmonary exercise test (CPET) to get the change of values of VE/VCO2 from 6th week(intervention ends) to 12th week(follow up ends)
Change of muscle strength from 1st week to 6th week | From 1st week to 6th week
  Use dynamometer to measure the changes of muscle strength(kg) from 1st week(intervention starts) to 6th week(intervention ends), including bilateral handgrip, elbow flexors (biceps) and knee extensors (quadriceps) for 3 times separately.The patient need to increase the strength to the highest level in 6 seconds and rest for 30 seconds.The highest value will be divided by the patient's body weight (kg/kg)
Change of muscle strength from 1st week to 12th week | From 1st week to 12th week
  Use dynamometer to measure the changes of muscle strength(kg) from 1st week(intervention starts) to 12th week(follow up ends), including bilateral handgrip, elbow flexors (biceps) and knee extensors (quadriceps) for 3 times separately.The patient need to increase the strength to the highest level in 6 seconds and rest for 30 seconds.The highest value will be divided by the patient's body weight (kg/kg)
Change of muscle strength from 6th week to 12th week | From 6th week to 12th week
  Use dynamometer to measure the changes of muscle strength(kg) from 6th week(intervention ends) to 12th week(follow up ends), including bilateral handgrip, elbow flexors (biceps) and knee extensors (quadriceps) for 3 times separately.The patient need to increase the strength to the highest level in 6 seconds and rest for 30 seconds.The highest value will be divided by the patient's body weight (kg/kg)
Change of 6-minute walk test from 1st week to 6th week | From 1st week to 6th week
  Measure the change of 6-minute walk test from 1st(intervention starts) week to 6th week(intervention ends).The patient walks in his/her own pace, as far as he/she can in 6 minutes at the 20-meter long straight path and the we will record the distance in meter.Stop when time's up or patient develops clinical symptoms.
Change of 6-minute walk test from 1st week to 12th week | From 1st week to 12th week
  Measure the change of 6-minute walk test from 1st(intervention starts) week to 12th week(follow up ends).The patient walks in his/her own pace, as far as he/she can in 6 minutes at the 20-meter long straight path and the we will record the distance in meter.Stop when time's up or patient develops clinical symptoms.
Change of 6-minute walk test from 6th week to 12th week | From 6th week to 12th week
  Measure the change of 6-minute walk test from 6th(intervention ends) week to 12th week(follow up ends).The patient walks in his/her own pace, as far as he/she can in 6 minutes at the 20-meter long straight path and the we will record the distance in meter.Stop when time's up or patient develops clinical symptoms.
Attendance rate in video group or booklet group | From 1st week to 6th week
  If the patient completes 70% or more of the intervention program by being analyzed from the record of RPE form, he/she will be recognize as being completed the intervention.Finally, we will count the number of the patients who completed the intervention to be divided by the number of totally patients in video/booklet group at 6th week.

SECONDARY OUTCOMES:
FEV1 | Baseline, 6 weeks later, and 12 weeks later
  Use spirometry to measure the values of FEV1 (%) for 3 times.The highest result will be recored.
FEV1/FVC | Baseline, 6 weeks later, and 12 weeks later
  Use spirometry to measure the values of FEV1/FVC for 3 times.The highest result will be recored.
Modified Medical Research Council (mMRC) | Baseline, 6 weeks later, and 12 weeks later
  Level of Modified Medical Research Council (mMRC)
COPD Assessment Test (CAT) | Baseline, 6 weeks later, and 12 weeks later
  Total score of COPD Assessment Test (CAT)
EuroQol-5 Dimensions-5 Levels (EQ-5D-5L) | Baseline, 6 weeks later, and 12 weeks later
  Score of EuroQol-5 Dimensions-5 Levels (EQ-5D-5L)
Clinical COPD Questionnaires (CCQ) | Baseline, 6 weeks later, and 12 weeks later
  Score of Clinical COPD Questionnaires (CCQ)

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hsia Hung, Ph.D, Study Chair — National Cheng-Kung University Hospital
Locations (1):
- National Cheng Kung University Hospital, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: No